CLINICAL TRIAL: NCT06360627
Title: Ultra Low Dose CT and Use of Iomeron 400 in PCD-CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022_D0008
Record Dates: First submitted 2023-02-27; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Radiation Exposure; Lung Embolism; Lung Cancer; Pneumonia
MeSH Terms: conditions — Pulmonary Embolism; Lung Neoplasms; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Dose (Other): Standard Low Dose CT
  Interventions: Radiation: Computed Tomography
- Ultra Low Dose (Other): Ultra Low Dose CT
  Interventions: Radiation: Computed Tomography

INTERVENTIONS:
Radiation: Computed Tomography — Computed Tomography CHEST

SUMMARY:
Evaluation of ultra low dose protocols and Iomeron 400 contrast in PCD-CT

ELIGIBILITY:
Inclusion Criteria:

* CT SCAN for pulmonary nodule detection/follow up
* CT SCAN for pneumonia detection/follow up

Exclusion Criteria:

* under 18
* BMI over 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose Reduction by new scanner | through study completion, an average of 1 year
  mSv per exam will be recorded. This value will be put in correlation to weight (Kg), height (cm) and BMI.
stable Image Quality in reduced dose scans | through study completion, an average of 1 year
  Recorded values compared in 2 populations-different contrast agents by using qualitative&quantitative methods Qualitative:diagnostic certainty, assessability of lung structure/lesions,diagnostic reliability,
  Quantitative:Assessment of tissue composition,diagnostic performance measurements Attenuation/sealing measurement (HU), signal-to-noise ratio (SNR), contrast-to-noise ratio ,size dimensions of lung structure/lesion in three dimensions in millimeters Tissue composition assessment diagnostic performance measurements (sensitivity, specificity, accuracy) diagnostic confidence: 1-4
  Theses measurements will be put in correlation to the scan dose (mSv) per patient, forming two groups with matched BMI (kg/m^2)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich - Diagnostic Radiology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No